CLINICAL TRIAL: NCT05200195
Title: Development and Validation of a Deep Learning Model for the Prediction of Hepatocellular Cancer Recurrence After Transplantation: The Time-Radiological Response- AlphafetoproteIN-Artificial Intelligence Model
Brief Title: Deep Learning Model for the Prediction of Post-LT HCC Recurrence
Acronym: TRAIN-AI
Status: Completed | Type: Observational
Sponsor: European Hepatocellular Cancer Liver Transplant Group (Other)
Responsible Party: Principal Investigator, Quirino Lai, Principal Investigator, European Hepatocellular Cancer Liver Transplant Group
Other Study IDs: #004
Record Dates: First submitted 2022-01-07; First posted 2022-01-20 (Actual); Last update posted 2022-06-30 (Actual); Status verified 2022-06

CONDITIONS: Liver Transplant Disorder; Liver Cancer; Recurrent Cancer
Keywords: artificial intelligence; deep learning; mathematical model
MeSH Terms: conditions — Liver Neoplasms; Recurrence | interventions — Liver Transplantation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- International Cohort Training Set: The Training Set of the International Cohort (N=3,670) was composed of the 80% (n=2936) HCC patients transplanted from 2000 to 2018 across 17 centers in Europe and Asia.
  Interventions: Procedure: Liver transplantation
- International Cohort Test Set: The Test Set of the International Cohort (N=3,670) was composed of the 20% (n=734) HCC patients transplanted from 2000 to 2018 across 17 centers in Europe and Asia.
  Interventions: Procedure: Liver transplantation
- Validation Cohort: The external Validation Cohort was composed of 356 HCC patients transplanted at the Columbia University, New York, during the period 2000-2018.
  Interventions: Procedure: Liver transplantation

INTERVENTIONS:
Procedure: Liver transplantation — Deceased or living donor liver transplantation for the cure of hepatocellular cancer on cirrhosis

SUMMARY:
Identifying patients at high risk for recurrence of hepatocellular carcinoma (HCC) after liver transplantation (LT) represents a challenging issue. The present study aims to develop and validate an accurate post-LT recurrence prediction calculator using the machine learning method.

DETAILED DESCRIPTION:
In 1996, the introduction of the Milan criteria (MC) strongly modified the selection process of hepatocellular cancer (HCC) patients waiting for liver transplantation (LT). Many attempts to widen MC have been proposed. Initially, exclusively morphology-based (nodules number and target lesion diameter) criteria were created. In the last years, extended criteria also based on biological parameters have been added. Among the most adopted biology-based features, the levels of different tumor markers, liver function parameters like the model for end-stage liver disease (MELD), the radiological response after neo-adjuvant therapies, and the length of waiting-time (WT) can be reported.

Unfortunately, all the proposed models showed suboptimal prediction abilities for the risk of post-LT recurrence. Such impairment was derived from the limitations of the standard statistical methods to account for many variables and their non-linear interactions. Therefore, developing a model based on Artificial Intelligence (AI) represents an attractive way to improve prediction ability.

Thus, the investigators hypothesize that an AI model focused on an accurate post-transplant HCC recurrence prediction should improve our ability to pre-operatively identify patients with different classes of risk for HCC recurrence after transplant.

This study aims to develop an AI-derived prediction model combining morphology and biology variables. A Training Set derived from an International Cohort was adopted for doing this. A Test Set derived from the same International Cohort and a Validation Cohort were adopted for the internal and external validation, respectively. A user-friendly web calculator was also developed.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive adult (≥18 years) patients enlisted and transplanted with the primary diagnosis of HCC during the period 2000-2018.

Exclusion Criteria:

* Patients with HCC diagnosed only at pathological examination (incidental HCC)
* Patients with mixed hepatocellular-cholangiocellular cancer misdiagnosed as HCC
* Patients with cholangiocellular cancer misdiagnosed as HCC
* Patients dying early after LT (≤ one month)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All the consecutive adult (≥18 years) patients enlisted and transplanted with the primary diagnosis of HCC during the period 2000-2018 in the 18 centers composing the International and the Validation Cohorts
Sampling Method: Probability Sample
Enrollment: 4026 (Actual)
Dates: Start 2020-01-15 (Actual); Primary Completion 2021-12-15 (Actual); Study Completion 2022-03-15 (Actual)

PRIMARY OUTCOMES:
Post-transplant HCC recurrence | 5 years from liver transplantation
  Intra- and/or extrahepatic recidivism of HCC after liver transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Quirino Lai, MD PhD, Principal Investigator — University of Roma La Sapienza
Locations (1):
- Quirino Lai, Rome, RM, Italy

IPD SHARING:
Plan to Share IPD: No